CLINICAL TRIAL: NCT01213498
Title: The Effects of Atorvastatin on the Nitric Oxide-system in Patients With Non-diabetic Nephropathy
Acronym: STAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Erling Bjerregaard Pedersen (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, professor, chief physician, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EBP-FHC-2010-2
Record Dates: First submitted 2010-09-19; First posted 2010-10-04 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Nephropathy; Cardiovascular Diseases
Keywords: Nephrology; Atorvastatin; L-NMMA; NO
MeSH Terms: conditions — Kidney Diseases; Cardiovascular Diseases | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Active Comparator)
  Interventions: Drug: Atorvastatin
- Unikalk (Placebo Comparator)
  Interventions: Drug: Unikalk

INTERVENTIONS:
Drug: Atorvastatin — Zarator, 80 mg pr. day for 5 days
  Other Names: Zarator
  Arms: Atorvastatin
Drug: Unikalk — 1 tablet Unikalk pr day for 5. days
  Arms: Unikalk

SUMMARY:
It has been documented that statin reduce mortality and morbidity in patients with cardiovascular disease. This effect can partly be related to a reduction in cholesterol levels in blood. Nitric oxide (NO) production is reduced in several chronic diseases such as nephropathy, diabetes and hypertension. The purpose of this study is to investigate the effect of Atorvastatin treatment on the NO-system measuring renal and cardiovascular variables in patients witk chronic kidney disease.

DETAILED DESCRIPTION:
Subjects will be examined on two examination days. 4 days prior to each examination day subjects are treated with either atorvastatin or placebo. During treatment periods subject are given a standardized diet.

On the examination days subject are given L-NMMA(L-NG-monomethyl Arginine citrate), a NO inhibitor, 6 mg bolus infusion followed by continuous 4 mg/kg/hr infusion for 1 hour. Renal function, central hemodynamic and vasoactive hormones are evaluated prior, during and after L-NMMA infusion.

Renal function is measured by renal clearance of 51Chromium-EDTA and urinary sodium, potassium and albumin concentration. Urinary excretion of protein from NCC, NKCC and ENaC will be measured to evaluate channel activity in the nephron.

Central blood pressure, pulse wave analysis, and augmentation index are measured using SphygmoCor® from Atcor.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* minimum 20 years
* Chronic Kidney disease
* Estimated GFR (eGFR) between 30 and 90 ml/min

Exclusion Criteria:

* Nephrotic Syndrome
* Diabetes mellitus
* Anamnestic or clinical signs of significant heart, lung, lever, kidney, thyroid and brain disease
* Neoplastic disease
* Alcohol abuse,
* Drug abuse
* Pregnancy or nursing
* Blood donation within a month before examination
* Hgb < 6,0

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Fractional excretion of sodium (FeNa) | 5 days treatment
  Fractional excretion of urinary sodium before, during and after L-NMMA infusion

SECONDARY OUTCOMES:
Systolic blood pressure | 5 days
Plasma renin concentration | 5 days
Arterial stiffness (Pulse wave velocity) | 5 days
Diastolic blood pressure | 5 day
Augmentation Index | 5 days
Urinary albumin excretion | 5 days
Urinary excretion of protein from sodium channels such as the NaCl cotransporter (NCC), the Na-K-Cl cotransporter (NKCC) and the epithelial sodium channel (ENaC) | 5 days
plasma aldosterone concentration | 5 days
Urinary Aquaporin 2(u-AQP2) excretion | 5 days
atrial natriuretic peptide (ANP) concentration | 5 days
Brain natriuretic peptide concentration | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medicinsk Forskning, Regionshospitalet Holstebro, Holstebro, Denmark

REFERENCES:
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702